CLINICAL TRIAL: NCT04701112
Title: Acute Hemodynamic Effects of His-bundle Pacing in Bi-Ventricular Pacing Non-responders (The HEPA-His Trial)
Brief Title: Acute Hemodynamic Effects of Pacing the His Bundle in Heart Failure
Acronym: HEPA-His
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic challenges
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Hepa-His trial
Record Dates: First submitted 2020-12-18; First posted 2021-01-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure, Systolic; Left Bundle Branch Block; Wide QRS Complex
Keywords: His Bundle pacing; Cardiac Resynchronization Therapy; Pacemaker
MeSH Terms: conditions — Heart Failure, Systolic; Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient is not aware of the pacing modality used for each measurement. The outcomes assessment will be performed blinded to pacing modality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- His-bundle pacing first (Experimental): AV sequential His-bundle pacing (or VVI pacing if in atrial fibrillation) via temporary right atrial and His-bundle electrodes.
  Then AV sequential Biventricular pacing via the patient's already implanted CRT device.
  Measurements of stroke volume, cardiac output, pressure in the right ventricle and pulmonary capillary wedge pressure, during rest and exercise. Simultaneous 12 lead ECG registration.
  Interventions: Device: Temporary His bundle pacing
- Biventricular pacing first (Active Comparator): AV sequential biventricular pacing (or VVI pacing if in atrial fibrillation) via the patient's already implanted CRT device. Then AV sequential or VVI His-bundle pacing via temporary right atrial and His-bundle electrodes.
  Measurements of stroke volume, cardiac output, pressure in the right ventricle and pulmonary capillary wedge pressure, during rest and exercise. Simultaneous 12 lead ECG registration.
  Interventions: Device: Temporary His bundle pacing

INTERVENTIONS:
Device: Temporary His bundle pacing — Temporary use of a Medtronic 3830 electrode placed in the region of His bundle, in combination with a Medtronic 5392 dual chamber external pacemaker and a temporary Edwards D200F7 Swan Ganz Pacing -catheter with atrial pacing capability.
  AV synchronous pacing (DDD 60/minute during rest and 120/minute during exercise, AV delay 150/180ms) will be performed using the atrial port (pacing catheter atrial electrodes) and ventricular port (His bundle electrode), or in the case of atrial fibrillation, only pacing the the His bundle in VVI mode 60/minute during rest and 120/minute during exercise.
  The Swan-Ganz will then be used for hemodynamic measurements during pacing. A Cardiotek ECG system will be used for simultaneous 12 lead ECG registration.

SUMMARY:
Cardiac resynchronization therapy (CRT) with biventricular pacing (BVP) is indicated for patients with low ejection fraction and persistent symptoms of heart failure despite medical therapy and a wide QRS-complex, preferably with a left bundle branch block. Unfortunately, up to 40 % receiving CRT do not respond with subjective improvement or improved left ventricular ejection fraction from the treatment.

There are few therapeutic alternatives in patients not responding to CRT with BVP, and the potential to improve cardiac function in these patients could make a large difference in terms of life quality and prognosis.

His-bundle pacing (HBP) can be a suitable alternative, but is likely not possible in all patients with failed CRT. Furthermore, upgrading to HBP does require a surgical procedure and therefore exposes the patients to risk of complications (e.g. infection of the device). Therefore, early identification of the patients who are likely to benefit from an upgrade to HBP would be beneficial.

This study aims to evaluate if patients with failed CRT treatment will benefit from hemodynamic improvement if they are treated with temporary HBP, without opening the device-pocket, and exposing the existing pacemaker-device to a risk of infection. A temporary pacemaker lead and pacing sheath will be used, and placed in the heart via a blood vessel on the right side of neck, using local anaesthesia. Acute effects on the pump function of the heart will be measured during rest and during supine bicycle test (the equivalent of moderate physical activity). Factors associated with a beneficial effect will be evaluated on a group basis.

If the individual patient experiences an improvement of cardiac function during the test, he/she will be offered an upgrade to HBP and a replacement of the existing device.

DETAILED DESCRIPTION:
Primary hypothesis:

His-bundle pacing will lead to a better stroke volume at rest compared to biventricular pacing.

Primary outcome measure:

Stroke-volume (ml) at rest assessed by invasive hemodynamic measurements with the thermodilution method using a Swan-Ganz catheter.

Recruitment:

Patients will be recruited from the dedicated CRT outpatient clinic at Skane University Hospital. This outpatient clinic evaluates all CRT recipients at 6 months after device implant. If the patient is then a "non-responder" by subjective and objective measures, it is unlikely that there will be any further benefit from the CRT device. Those patients fulfilling the inclusion criteria but not the exclusion criteria will therefore be invited to participate in the study. Written information will be provided to all patients prior to informed consent is signed.

Procedure:

All patients will undergo a temporary His-bundle stimulation and hemodynamic evaluation. The procedure takes place at the dedicated laboratory for advanced hemodynamic evaluation at Skåne University Hospital in Lund. The first option for vascular access is the right external jugular vein. Under sterile conditions, ultrasound guided venous puncture will be performed, using standard Seldinger technique. A 7F catheter (Medtronic C315) will then be placed over a long guidewire, and used to direct a dedicated pacemaker lead (Medtronic Select Secure 3830) to the His bundle. In case of technical difficulties, a steerable 9F catheter will be used instead (Medtronic C304 deflectable). If HBP is not possible using jugular access, an alternate access via the right femoral vein may be used instead. If the femoral vein is used, only resting measurements will be performed, since it is not possible to thread on the supine bike with a catheter in situ via the femoral vein. In parallel, in a short 8F introducer, a 7F multilumen Swan Ganz catheter will be placed over a long guidewire, and advanced to the left or right pulmonary artery. The catheter will then be wedged in a pulmonary segmental artery to obtain left atrial pressure curves.

The pacing lead will be connected to an electrophysiology 12-lead ECG system with capability of pacing and continuous ECG registration of external and intracardiac signals. His bundle potential will be identified probing the correct anatomical area with the electrode, and subsequently the pacing properties of the electrode will be tested. If the pacing properties result in selective (or subsidiary non-selective) his bundle capture, the electrode will be secured in place by 2-3 careful rotations of the entire electrode. The goal is to achieve a stable position with minimal risk of damaging the conduction system by trauma. Since the patients are paced using the CRT device anyway, trauma to the conduction system will not be deleterious, but it may hamper the ability to place a permanent HBP lead at a later stage, if that is indicated. When stable pacing conditions are in place, the stimulation program will be initiated. Depending on randomization results, the intrinsic CRT system or the temporary His-lead will be used for pacing. Pacing and sensing in the right atrium will be achieved using atrial electrodes on the outside of the Swan Ganz catheter.

The patients are randomized to wither Biventricular pacing first or HBP first. The pacing program involves both pacing at rest and pacing during sub maximal exercise test (supine bicycle test). Each pacing step is sustained at steady state for at least 2 minutes prior to measurement of intracardiac pressures, cardiac output and stroke volume calculations. After the pacing protocol is finished, the catheters are withdrawn and the site of venopuncture is manually compressed during 5 minutes. The patients are then observed during 2 hours, before discharge and completion of the study.

A hemodynamic optimization will be performed regarding device settings for all patients. Patients who have a positive hemodynamic response to HBP, compared to CRT pacing, will at a follow-up stage be offered an upgrade to permanent HBP.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Native QRS-duration >130 ms and a left bundle branch block or previous His-ablation
* Heart failure in New York Heart Association functional class II-IV
* Echocardiographic non-responder to ongoing CRT defined as <15% reduction in LVESV compared to pre-CRT examination
* Clinical non-responder to ongoing CRT, defined as lack of subjective improvement after CRT
* Signed informed consent

Exclusion Criteria:

* Known access site problems in vena jugularis interna dx or sin
* Not able to perform supine cycling
* Presence of severe tricuspid regurgitation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Change in stroke volume (ml) at rest, between Biventricular pacing compared to His bundle pacing | During procedure
  Stroke volume will be measured using the thermodilution method, and paired T-test will be used to evaluate the change in stroke volume between the different pacing modes.

SECONDARY OUTCOMES:
Change in stroke volume (ml) at sub-maximal exercise, between Biventricular pacing compared to His bundle pacing | During procedure
  Stroke volume (ml) measured by the thermodilution method.
Change in Cardiac output (l/min) at rest, between Biventricular pacing compared to His bundle pacing | During procedure
  Cardiac output (l/min) at rest assessed by invasive hemodynamic measurements with the thermodilution method.
Change in cardiac output (l/min) at submaximal exercise, between Biventricular pacing compared to His bundle pacing | During procedure
  Cardiac output (l/min) at sub-maximal exercise assessed by invasive hemodynamic measurements with the thermodilution method using a Swan-Ganz catheter.
Change in stroke work index (mmHg x ml/m2) at rest, between Biventricular pacing compared to His bundle pacing | During procedure
  Calculation of stroke work index based on invasive measurements
Change in stroke work index (mmHg x ml/m2) at sub-maximal exercise, between Biventricular pacing compared to His bundle pacing | During procedure
  Calculation of stroke work index based on invasive measurements
Change in QRS vector area, between Biventricular pacing compared to His bundle pacing | During procedure
  Change in high resolution digital ECG recording of QRS vector area

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events, defined as pneumothorax or pericardial effusion. | From start of procedure to 2 hours post-procedure
  If the patient develops symptoms of respiratory discomfort and/or blood pressure drop ≥10mmHg during or within 2 hours after the procedure, evaluation by chest X-ray and echocardiography will be performed. Presence of pneumothorax or pericardial effusion will be documented as adverse events.
Incidence of Treatment-Emergent Adverse Events, defined as local access site bleeding. | From start of procedure to 2 hours post-procedure
  If there is bleeding that requires compression >10minutes it will be recorded as an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Braun, MD PhD, Principal Investigator — Region Skane, Lund University; Rasmus Borgquist, MD PhD, Principal Investigator — Region Skane, Lund University
Locations (1):
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No